CLINICAL TRIAL: NCT00548886
Title: Low-dose Epinephrine Infusion Tests in Adolescent and Pediatric Patients
Acronym: LEAP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: Emory University (Other)
Collaborators: Children's Healthcare of Atlanta (Other)
Responsible Party: Principal Investigator, Peter Fischbach, Associate Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB00008105
Record Dates: First submitted 2007-10-22; First posted 2007-10-24 (Estimated); Results first posted 2015-03-06 (Estimated); Last update posted 2017-12-06 (Actual); Status verified 2017-11

CONDITIONS: Congenital Disorders
Keywords: QT Prolongation; QT Interval; Epinephrine; Stress test
MeSH Terms: conditions — Congenital, Hereditary, and Neonatal Diseases and Abnormalities; Long QT Syndrome | interventions — Epinephrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Epinephrine (Experimental): Healthy pediatric subjects will receive epinephrine. Epinephrine infusion will begin at 0.025 ug/kg/minute, for ten minutes.The epinephrine infusion will then be increased to 0.05 ug/kg/minute for five minutes. The epinephrine infusion will then be increased to a maximal dose of 0.1 ug/kg/minute for five minutes. The epinephrine infusion is then discontinued.
  Interventions: Drug: Epinephrine

INTERVENTIONS:
Drug: Epinephrine — We will follow the protocol outlined by Ackerman et al. known as the Mayo protocol4 which is currently used routinely in our electrophysiology laboratory. Epinephrine infusion will begin at 0.025 ug/kg/minute, for ten minutes and a twelve-lead electrocardiogram is obtained at time=0 minutes, 5 minutes, and 10 minutes. The epinephrine infusion will then be increased to 0.05 ug/kg/minute for five minutes and the electrocardiogram repeated. The epinephrine infusion will then be increased to a maximal dose of 0.1 ug/kg/minute for five minutes and electrocardiogram obtained. The epinephrine infusion is then discontinued and measurements are obtained at five minutes and ten minutes after stopping the epinephrine infusion. The total time of procedure will be 35 minutes.
  Other Names: adrenaline

SUMMARY:
Long QT syndrome (LQTS)is a cardiac disorder that may lead to ventricular arrythmias and culminate in syncope and/or possible death.

Recently, researchers have developed a way of discovering patients with LQTS by using low doses of epinephrine by a continuous, intravenous infusion in adults. Epinephrine, or adrenaline, is produced by our bodies in times of stress. By producing adrenaline, your body allows itself to adapt to its stressful environment and take appropriate actions (i.e. fight or flight response). By simulating this response with very small amounts of epinephrine, researchers have shown prolongation of the QT interval does not occur in normal healthy adults. However, adults with confirmed LQTS Type 1 (LQTS-1) will prolong their QT interval when given low dose epinephrine. Therefore, this test can act as a safe means of identifying adults with LQTS-1 who do not have prolonged QT intervals on their resting EKGs.

However, LQTS is not just a disease of adults, it affects children as well. Currently the standard of care is to obtain resting EKGs on our pediatric patients which can miss those patients with concealed LQTS. Those patients, who are old enough, can undergo exercise testing. Yet this leaves young children unable to run on a treadmill without a diagnostic test.

Hypothesis: The low-dose epinephrine infusion stress test does not cause prolongation of the QT interval in an electrophysiologically normal healthy pediatric population.

DETAILED DESCRIPTION:
This study will involve asking fifty children coming to the hospital for their standard of care procedure to treat a separate cardiac condition to participate. Patients approached will already have an intravenous line in place for their procedure. After consent and assent as necessary are obtained, the patient be brought to a separate room for the low-dose epinephrine infusion trial. The patient will lie down on a table, be hooked up to an EKG machine and the infusion will start. The amount of epinephrine actually infused is based on the weight of the patient but is substantially less than the dose received from an epinephrine auto-injection for anaphylaxis. After about 40 minutes, the trial will be completed and the patient may return to the waiting room for their original procedure. We have performed this test on a number of pediatric patients suspected of having LQTS with promising results and with little to no side effects. The patient will be awake for the procedure and will be able to verbalize concerns or complaints. A pediatric electrophysiologist and nurse will be present throughout the entire procedure.

The purpose of this study is to determine if children who are infused with low amounts of epinephrine will also maintain their normal QT interval as it does with healthy adults. This study would hope to prove that low-dose epinephrine infusion trials can serve as a way of identifying children with LQTS so that they may be effectively treated and potentially have their lives saved.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ages 3-18 years
2. Patients undergoing device closure of an atrial septal defect in the cardiac catheterization lab
3. normal electrocardiogram without prolonged absolute or corrected QT interval(less than 440 msec)

Exclusion Criteria:

1. Patients with a history of any other structural or acquired heart disease besides the atrial septal defect.
2. Patient with a family history of sudden cardiac death, or personal history of syncope.
3. Patient on alpha or beta-blocking medications.
4. Pregnancy.

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 7 (Actual)
Dates: Start 2008-02; Primary Completion 2012-01 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Fischbach, MD, MA, Principal Investigator — Emory University
Locations (1):
- Children's Healthcare of Atlanta, Atlanta, Georgia, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects recruited from Children's Healthcare of Atlanta (CHOA) February 2008 through January 2012
Period: Overall Study
Arm/Group | Epinephrine
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Epinephrine
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 7
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 5

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With a Positive Result in Absolute QT Interval
Description: QT interval refers to the time interval on the standard electrocardiogram from the beginning of the QRS complex to the end of the T wave. Each participant had four QT intervals measured at each timepoint and the average was calculated for each patient at each timepoint for an absolute QT interval. Lengthening of the absolute QT interval greater than 30 milliseconds on low dose epinephrine infusion would be considered a positive result.
Time Frame: 35 minutes
Population: Data not analyzed due to study termination
Arm/Group | Epinephrine
Number analyzed (Participants) | 0

2. Secondary Outcome: Determine Interobserver Variability When Measuring QT Intervals
Description: Two pediatric electrophysiologists were given photocopies of rhythm strips obtained from the electrocardiograms and the electrophysiologists will then take four separate measurements of the QT interval from each rhythm strip. Interobserver variability was measured between the two electrophysiologists and their measurements on the same rhythm strip. False positive results will be based on measurement error.
Time Frame: During enrollment period
Population: Interobserver variability was not performed due to study termination
Arm/Group | Epinephrine
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Epinephrine
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 0/7

LIMITATIONS AND CAVEATS:
Slow enrollment lead to an early termination of the study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes